CLINICAL TRIAL: NCT01852487
Title: Effect of Pumpkin Seed Oil on Hair Growth in Men With Androgenetic Alopecia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dream Plus (Industry)
Responsible Party: Principal Investigator, Young Hye Cho, Professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pumpkin0912
Record Dates: First submitted 2013-05-09; First posted 2013-05-13 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: Androgenic Alopecia
Keywords: Pumpkin seed oil; Hair growth; Men
MeSH Terms: conditions — Alopecia; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Pumpkin Seed Oil (Active Comparator): 400mg/ day during 6 months
  Interventions: Dietary Supplement: 400mg /day during 6 months
- sweet potato starch (Placebo Comparator): 400mg/day during 6months

INTERVENTIONS:
Dietary Supplement: 400mg /day during 6 months
  Arms: Pumpkin Seed Oil

SUMMARY:
Androgenic alopecia is the most common cause of hair loss in men. Finasteride and minoxidil are available in treatment of androgenetic alopecia, although the former causes decreased libido or ejaculate volume, erectile dysfunction, the latter causes scaling, itching of the scalp. Recently, Pulpkin Seed Oil shows some improved clinical efficacy on scalp hair growth in men with androgenetic alopecia, but there is no evidence to support this.

The investigators conducted a randomized, double-blind, placebo-controlled efficacy and tolerability trial of Pumpkin seed oil (400mg/day)therapy in male patients with androgenetic alopecia.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years of age
* Androgenetic alopecia of Norwood-Hamilton scale grade II-V

Exclusion Criteria:

* Severe medical problems including renal problems, prostate diseases, diabetes mellitus o
* Patients who took any medicine which can affect the hair growth in recent 3 months.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
investigator assessment score using photographs of scalp hair | at weeks 12 and 24

SECONDARY OUTCOMES:
patient self-assessment scores | at weeks 12 and 24

OTHER OUTCOMES:
hair analysis using phototrichogram | at weeks 12 and 24

CONTACTS AND LOCATIONS:
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do, South Korea